CLINICAL TRIAL: NCT02054572
Title: An Open-label, Single-dose Study to Evaluate the Pharmacokinetics, Biotransformation and Excretion of [¹⁴C]AMG 416 in Patients With End Stage Renal Disease Receiving Dialysis
Brief Title: Pharmacokinetics and Excretion of [¹⁴C]Etelcalcetide (AMG 416) in Patients With End Stage Renal Disease (ESRD) Receiving Dialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20130147
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Secondary Hyperparathyroidism in Patients With ESRD on Hemodialysis
Keywords: AMG 416, ESRD, hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [¹⁴C]Etelcalcetide (Experimental): Participants received a single dose of 10 mg radiolabelled etelcalcetide administered by intravenous (IV) bolus injection at the end of hemodialysis on day 1.
  Interventions: Drug: [¹⁴C]Etelcalcetide

INTERVENTIONS:
Drug: [¹⁴C]Etelcalcetide — 750 nCi of [¹⁴C]etelcalcetide formulated as a single 10 mg dose of etelcaletide in 2 mL liquid solution for bolus intravenous (IV) administration at the end of hemodialysis.
  Other Names: AMG 416; Parsabiv™

SUMMARY:
The primary objectives of this study were to determine the rate, extent, and routes of radioactivity excretion of [¹⁴C]etelcalcetide in feces, dialysate, and urine over time and to measure radioactivity concentrations in whole blood and plasma over time.

DETAILED DESCRIPTION:
Six adult male or female patients with end stage renal disease requiring hemodialysis will be enrolled to receive 750 nCi of [¹⁴C]-labeled etelcalcetide formulated in 10 mg etelcalcetide administered as a single 2 mL intravenous dose at the end of hemodialysis.

Participants will spend the first approximately 12 days in confinement at the clinic (day -1 until completion of day 11 study procedures). Blood samples, and complete collections of dialysate, dialysis membrane (as necessary), urine (as available), and feces will be analyzed for radioactivity content by accelerator mass spectrometry (AMS). Following the confinement period, participants will return to the site on an outpatient basis in accordance to their routine dialysis sessions up to day 39. Blood and dialysate samples and dialysis membranes will be collected at specified times during the outpatient visit period.

Participants may be asked to return so the site for the Extended Pharmacokinetic Collection Period. During the Extended Pharmacokinetic Collection Period, participants will return to the site for 3 consecutive hemodialysis sessions (Collection Period 1) and then again approximately one month later, for an additional 3 consecutive hemodialysis sessions (Collection Period 2).

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures.
* Male or female subject ≥ 18 years of age at the time of screening, with end stage renal disease receiving hemodialysis;
* Body mass index is between 18 and 38 kg/m², inclusive;
* Corrected calcium (calculated) level is > 8.3 mg/dL and intact parathyroid hormone (PTH) level is between 300 - 1200, inclusive; all other laboratory tests within clinically acceptable range to the investigator and sponsor at screening;
* Female subjects must be of non-reproductive potential (ie, postmenopausal by history - no menses for 1 year and follicle-stimulating hormone (FSH) level consistent with postmenopausal status; OR history of hysterectomy; OR history of bilateral tubal ligation);
* Negative screen for potential drugs of abuse at screening, unless positive result is expected based on approved concomitant medications;
* Negative alcohol test at screening;
* Subject has functioning permanent dialysis access via fistula, hemodialysis (HD) catheter, or arteriovenous (AV) graft;
* Subject must be receiving hemodialysis 3 times weekly for at least 1 year prior to day -1 (or is confirmed to be anuric based on historical and clinical assessment if on hemodialysis for less than one year), and have adequate hemodialysis with a delivered Kt/V ≥ 1.2 or urea reduction ratio (URR) ≥ 65% within 4 weeks to screening. The subject's routine hemodialysis session must be of 3-4.5 hours in duration, inclusive;
* Subject has stable dialysis prescription and this prescription is not anticipated to change significantly during the course of the study.

Exclusion Criteria:

* Female subjects who are lactating/breastfeeding or who plan to breastfeed while on study through 3 months after receiving the dose of study drug;
* Females with a positive pregnancy test at screening;
* Positive for human immunodeficiency virus (HIV) at screening or known diagnosis of acquired immune deficiency syndrome (AIDS);
* Positive Hepatitis B Surface Antigen (HepBsAg) at screening (indicative of chronic Hepatitis B);
* Positive for Hepatitis C virus ribonucleic acid (RNA) by polymerase chain reaction (PCR) at screening (indicative of active hepatitis C - screening is generally done by hepatitis C antibody (HepCAb), followed by hepatitis C virus RNA by PCR if HepCAb is positive);
* Previous administration of AMG 416;
* Previous administration of any [¹⁴C] labeled drug substance within 1 year before study drug administration;
* Subject has received cinacalcet within the 30 days prior to study drug administration (treatment with cinacalcet is prohibited during the study);
* Subject has known sensitivity to any of the products or components to be administered during dosing;
* Use of concomitant medication other than that used in the management of end stage renal disease and its expected comorbidities that could in the opinion of the investigator or Amgen medical monitor interfere with the safety of subjects or interpretation of study results;
* Known illicit drug abuse within 12 months of day -1;
* Unwilling or unable to limit alcohol consumption throughout the course of the study;
* Alcohol is limited to no more than 2 units per day during the outpatient period of the study through completion of day 39. A standard unit is equivalent to 12 ounces of regular beer, 8-9 ounces of malt liquor, 5 ounces of wine, or 1.5 ounces of 80 proof distilled spirits;
* Receiving or has received any investigational drug (or is currently using an investigational device) within the 30 days before receiving study drug, or at least 10 times the respective elimination half-life (whichever is longer);
* Subject has lost 500 mL or more of blood or plasma within 8 weeks of study drug administration or during the study period;
* Subjects with hemodynamic instability during hemodialysis;
* Anticipated or scheduled kidney transplant during the study period
* Subject has an unstable medical condition based on medical history, physical examination, and routine laboratory tests, or is otherwise unstable in the judgment of the Investigator;
* Subject has an active infection at screening or day -1, or a history of any illness that, in the opinion of the Investigator, might confound the results of the study or pose additional risk to the subject;
* History of malignancy (within 5 years before day -1) of any type, other than surgically excised non-melanomatous skin cancers;
* Subject's 12-lead electrocardiogram (ECG) at screening suggests unstable arrhythmia or other cardiac abnormality that could place the subject at increased risk, based upon the Investigator's opinion
* Subject has poorly controlled hypertension;
* Subject has a history of symptomatic ventricular dysrhythmias or Torsades de Pointes;
* Subject has a history within the past 6 months of angina pectoris with symptoms that occur at rest or minimal activity or a history of congestive heart failure (New York Heart Association Classification III or IV);
* Subject has a history of myocardial infarction, coronary angioplasty, or coronary arterial bypass grafting within the past 6 months prior to screening;
* Subject is receiving treatment for a seizure disorder or has a history of a seizure within the last 12 months prior to screening;
* Subject has had major surgery (excluding minor surgery and hemodialysis access repair) within the last 8 weeks prior to screening;
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and Investigator's knowledge;
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02-07 (Actual); Primary Completion 2014-04-15 (Actual); Study Completion 2014-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- DaVita Clinical Research Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Wu L, Melhem M, Subramanian R, Wu B. Drug disposition model of radiolabeled etelcalcetide in patients with chronic kidney disease and secondary hyperparathyroidism on hemodialysis. J Pharmacokinet Pharmacodyn. 2017 Feb;44(1):43-53. doi: 10.1007/s10928-016-9503-z. Epub 2017 Jan 6. PMID 28063122
- [Background] Wu B, Melhem M, Subramanian R, Chen P, Jaramilla Sloey B, Fouqueray B, Hock MB, Skiles GL, Chow AT, Lee E. Clinical Pharmacokinetics and Pharmacodynamics of Etelcalcetide, a Novel Calcimimetic for Treatment of Secondary Hyperparathyroidism in Patients With Chronic Kidney Disease on Hemodialysis. J Clin Pharmacol. 2018 Jun;58(6):717-726. doi: 10.1002/jcph.1090. Epub 2018 Mar 13. PMID 29534286
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States from 07 February 2014 to 15 August 2014.
Period: Overall Study
Arm/Group | [¹⁴C]Etelcalcetide
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black (or African American) | 5
  Native Hawaiian or Other Pacific Islander | 0
  White | 1

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Excretion of Radioactivity
Description: The total radioactivity in excreta (urine and feces) or dialysate and dialysis membrane is expressed as a percentage of the total radioactive [¹⁴C] administered (dose). Total radioactive counts in dialysate, dialyzer, feces, and urine were determined by accelerator mass spectrometry (AMS). Radioactivity excreted during non-sampled days was estimated by interpolation and extrapolation of the measured data.
Time Frame: Day 1 to day 176
Population: Participants who received any amount of [¹⁴C]etelcalcetide with available excretion data
Measure: Mean (Standard Deviation); unit: Percentage of administered dose
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 4
Percentage of administered dose
  Dialysate (Measured) | 35.29 (4.17)
  Dialysate (Estimated) | 24.26 (2.71)
  Urine (Measured) | 0.75 (1.13)
  Urine (Estimated) | 2.40 (3.79)
  Feces (Measured) | 1.17 (0.13)
  Feces (Estimated) | 3.34 (0.57)
  Total | 67.19 (1.37)

2. Primary Outcome: Time to Maximum Observed Concentration (Tmax) of [¹⁴C]Etelcalcetide-derived Radioactivity in Plasma
Description: Total radioactive counts in plasma was determined by accelerator mass spectrometry (AMS).
Time Frame: Samples were collected from pre-dose on day 1 to day 39; additional samples were collected at 3 consecutive hemodialysis sessions from days 129 -148 and approximately 1 month later at an additional 3 consecutive hemodialysis sessions from days 157-176.
Population: Participants who received any part of the [¹⁴C]etelcalcetide dose and had measurable concentrations in at least 1 sample were included in the analysis.
Measure: Median (Full Range); unit: minutes
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
minutes | 10 [10 to 12]

3. Primary Outcome: Maximum Observed Concentration (Cmax) of [¹⁴C]Etelcalcetide-derived Radioactivity in Plasma
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng-eq/mL
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
ng-eq/mL | 697 (207) [10 to 12]

4. Primary Outcome: Time to Last Observed Plasma Concentration of [¹⁴C]Etelcalcetide-derived Radioactivity in Plasma
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
days | 164 [37.6 to 174]

5. Primary Outcome: Last Observed Plasma Concentration (Clast) of [¹⁴C]Etelcalcetide-derived Radioactivity in Plasma
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: ng-eq/mL
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
ng-eq/mL | 3.01 [2.06 to 24.7]

6. Primary Outcome: Apparent Terminal Half-life (T½) of [¹⁴C]Etelcalcetide-derived Radioactivity in Plasma
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
days | 35.9 (2.99) [10 to 12]

7. Primary Outcome: Area Under the Curve From Time Zero to 3 Days Post-dose (AUC3d) of [¹⁴C]Etelcalcetide-derived Radioactivity in Plasma
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: day*ng-eq/mL
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
day*ng-eq/mL | 585 (98.8) [10 to 12]

8. Primary Outcome: Area Under the Curve From Time Zero to 10 Days Post-dose (AUC10d) of [¹⁴C]Etelcalcetide-derived Radioactivity in Plasma
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: day*ng-eq/mL
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
day*ng-eq/mL | 1220 (172) [10 to 12]

9. Primary Outcome: Area Under the Arterial Plasma Concentration-time Curve Obtained During Hemodialysis on Day 4 for Etelcalcetide
Description: Etelcalcetide plasma concentrations were determined by liquid chromatography-tandem mass spectrometry (LC-MS/MS).
Time Frame: Day 4 within 10 minutes after the start of hemodialysis, at 2 hours after the start of hemodialysis, and within 10 minutes before the end of hemodialysis.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
ng*day/mL | 1.79 (0.467) [10 to 12]

10. Primary Outcome: Area Under the Venous Plasma Concentration-time Curve Obtained During Hemodialysis on Day 4 for Etelcalcetide
Description: Etelcalcetide plasma concentrations were determined by liquid chromatography-tandem mass spectrometry (LC-MS/MS).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
ng*day/mL | 1.09 (0.264) [10 to 12]

11. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Etelcalcetide
Description: Etelcalcetide plasma concentrations were determined by liquid chromatography-tandem mass spectrometry (LC-MS/MS).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: minutes
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
minutes | 10 [10 to 11]

12. Secondary Outcome: Maximum Observed Concentration (Cmax) of Etelcalcetide
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
ng/mL | 347 (69.5) [10 to 12]

13. Secondary Outcome: Time to Last Observed Plasma Concentration of Etelcalcetide
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
days | 37.8 [37.6 to 145]

14. Secondary Outcome: Last Observed Plasma Concentration (Clast) of Etelcalcetide
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
ng/mL | 2.50 [0.210 to 2.80]

15. Secondary Outcome: Area Under the Curve From Time Zero to 3 Days Post-dose (AUC3d) of Etelcalcetide
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
day*ng/mL | 81.6 (8.41) [10 to 12]

16. Secondary Outcome: Area Under the Curve From Time Zero to 10 Days Post-dose (AUC10d) of Etelcalcetide
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
day*ng/mL | 160 (16.9) [10 to 12]

17. Secondary Outcome: Hemodialysis Clearance of Etelcalcetide During Hemodialysis on Day 4
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
mL/hr | 7660 (1380)

18. Secondary Outcome: Hemodialysis Extraction Ratio for Etelcalcetide During Hemodialysis on Day 4
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
ratio | 0.385 (0.0679)

19. Secondary Outcome: Number of Participants With Adverse Events
Description: A treatment-related adverse event (TRAE) is any adverse event (AE) that per investigator review has a reasonable possibility of being caused by the investigational product.
Time Frame: From first dose of etelcalcetide to day 39
Population: Participants who received any amount of [¹⁴C]etalcalcetide
Measure: Number; unit: participants
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
participants
  Any adverse event (AE) | 5
  Serious adverse events | 1
  AE leading to discontinuation of etelcalcetide | 0
  Fatal adverse events | 0
  Treatment-related adverse events (TRAEs) | 2
  Treatment-related serious adverse events | 0
  TRAE leading to discontinuation of etelcalcetide | 0
  Fatal treatment-related adverse events | 0

20. Secondary Outcome: Number of Participants With Anti-etelcalcetide Antibodies
Description: The presence of anti-etelcalcetide antibodies was assessed and confirmed using a dual-flow cell biosensor immunoassay at baseline (day -1) and at the end of study visit (day 39).
Time Frame: Day -1 and day 39
Population: Participants who received any amount of [¹⁴C]etalcalcetide
Measure: Number; unit: participants
Arm/Group | [¹⁴C]Etelcalcetide
Number analyzed (Participants) | 6
participants
  Pre-existing antibody incidence (Day -1) | 0
  Developing antibody incidence (Day 39) | 0

ADVERSE EVENTS:
Time Frame: From first dose of etelcalcetide to day 39.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- [¹⁴C]Etelcalcetide: Participants received a single dose of 10 mg radiolabelled etelcalcetide administered by IV bolus at the end of hemodialysis on day 1.
Arm/Group | [¹⁴C]Etelcalcetide
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [¹⁴C]Etelcalcetide (N=6)
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | [¹⁴C]Etelcalcetide (N=6)
Constipation (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.